CLINICAL TRIAL: NCT01825213
Title: Stratification of Patients With Chronic Liver Disease Using Multi Spectral CT
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Dushyant V. Sahani, Director of CT, Associate Professor of Radiology Harvard Medical School, Massachusetts General Hospital
Other Study IDs: 2013P000042
Record Dates: First submitted 2013-04-02; First posted 2013-04-05 (Estimated); Last update posted 2017-04-17 (Actual); Status verified 2017-01

CONDITIONS: Chronic Liver Disease; HepatoCellular Carcinoma; Liver Fibrosis
Keywords: Liver disease; Multi Spectral CT
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Cirrhosis; Liver Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Multispectral CT of the liver: Images of lesions and liver will be compared to histology.
  Interventions: Device: Multispectral CT of the liver

INTERVENTIONS:
Device: Multispectral CT of the liver — Analysis of the background liver and liver lesions will be performed on Multi Spectral CT images and compared to histology.
  Other Names: Discovery CT 750 HD, K120833

SUMMARY:
The purpose of this study is to evaluate the feasibility to stratify liver fibrosis in patients with chronic liver disease through non-invasive, spectral CT.

DETAILED DESCRIPTION:
This is a retrospective study, in which a FDA approved imaging device (spectral CT scanner) currently used for several clinical applications will be evaluated for feasibility of studying chronic liver disease (this application has not yet been validated).

Tomographic imaging has assumed a fundamental role in patients with Chronic Liver Disease (CLD) to screen patients for hepatocellular carcinoma (HCC), and, is increasingly being explored as a noninvasive alternative for characterizing liver fibrosis. The overarching goal of this study is to improve noninvasive characterization of liver fibrosis through spectral CT.

Hypothesis: concentration of iodine-based contrast agent in the liver parenchyma during the delayed phase, as measured with spectral CT imaging, increases monotonically with Ishak fibrosis score obtained from liver biopsy. This hypothesis is supported by the literature and our preliminary data, described in the references section (Lamb et al. 2015).

We will evaluate multiphase spectral CT images consisting of the arterial phase, 2-minute delayed phase, and 5-minute delayed phase. Fibrosis will be assessed on both delayed phase images, where it is assumed that any remaining contrast agent, in the liver, is due to the presence of fibrosis. This type of multiphase protocol can still be used to image CLD patients with spectral CT for HCC detection and, thus, will not interfere with liver lesion workup and evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient with chronic liver disease undergoing CT scan for/suspicion of hepatocellular carcinoma.
* Patients should be scheduled for/or should have obtained a multiphasic MRI of the liver.

Exclusion Criteria:

* Patients < 18 years old.
* History of allergy to intravenous contrast.
* Patients at risk for contrast-induced-nephropathy,
* Pregnant patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients with newly stablished diagnosis of hepatocellular carcinoma complying with selection criteria for liver transplantation and/or biopsy.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2013-11; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Detection of hepatocellular carcinoma on Multi Spectral CT | confirmation with focal biopsy and or/contrast-enhanced MRI of the liver acquired within 6 months prior to the multi spectral CT scan.

CONTACTS AND LOCATIONS:
Overall Officials: Dushyant V Sahani, MD, Principal Investigator — Director of CT, Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital,, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang G, Butler A, Yu H, Campbell M. Guest editorial. Special issue on spectral CT. IEEE Trans Med Imaging. 2015 Mar;34(3):693-6. doi: 10.1109/tmi.2015.2404591. No abstract available. PMID 25893236
- [Background] Zhao W, Niu T, Xing L, Xie Y, Xiong G, Elmore K, Zhu J, Wang L, Min JK. Using edge-preserving algorithm with non-local mean for significantly improved image-domain material decomposition in dual-energy CT. Phys Med Biol. 2016 Feb 7;61(3):1332-51. doi: 10.1088/0031-9155/61/3/1332. PMID 26796948
- [Background] Breguet R, Ronot M, Goossens N, Hansen C, Giostra E, Majno P, Becker CD, Spahr L, Terraz S. Liver volume is a prognostic indicator for clinical outcome of patients with alcoholic hepatitis. Abdom Radiol (NY). 2017 Feb;42(2):460-467. doi: 10.1007/s00261-016-0892-7. PMID 27604894
- [Background] Lestra T, Mule S, Millet I, Carsin-Vu A, Taourel P, Hoeffel C. Applications of dual energy computed tomography in abdominal imaging. Diagn Interv Imaging. 2016 Jun;97(6):593-603. doi: 10.1016/j.diii.2015.11.018. Epub 2016 Mar 15. PMID 26993967
- [Background] Patino M, Prochowski A, Agrawal MD, Simeone FJ, Gupta R, Hahn PF, Sahani DV. Material Separation Using Dual-Energy CT: Current and Emerging Applications. Radiographics. 2016 Jul-Aug;36(4):1087-105. doi: 10.1148/rg.2016150220. PMID 27399237
- [Background] Daginawala N, Li B, Buch K, Yu H, Tischler B, Qureshi MM, Soto JA, Anderson S. Using texture analyses of contrast enhanced CT to assess hepatic fibrosis. Eur J Radiol. 2016 Mar;85(3):511-7. doi: 10.1016/j.ejrad.2015.12.009. Epub 2015 Dec 17. PMID 26860661
- [Background] De Cecco CN, Boll DT, Bolus DN, Foley WD, Kaza RK, Morgan DE, Rofsky NM, Sahani DV, Schoepf UJ, Shuman WP, Siegel MJ, Vrtiska TJ, Yeh BM, Berland LL. White Paper of the Society of Computed Body Tomography and Magnetic Resonance on Dual-Energy CT, Part 4: Abdominal and Pelvic Applications. J Comput Assist Tomogr. 2017 Jan;41(1):8-14. doi: 10.1097/RCT.0000000000000546. PMID 27824670
- Available data/document: Peer reviewed article: PMID: 25181365 — http://ieeexplore.ieee.org/document/6887313/?arnumber=6887313